CLINICAL TRIAL: NCT06798571
Title: The Influence of Estrogen on the Thermoregulatory Responses to Heat Stress in Pre and Postmenopausal Women
Brief Title: Role of Menopause in Thermoregulation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, W. Larry Kenney, Professor, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Study 25435
Record Dates: First submitted 2025-01-15; First posted 2025-01-29 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Menopause; Aging
Keywords: Thermoregulation; Heat Stress
MeSH Terms: conditions — Heat Stress Disorders | interventions — elagolix; Ortho Evra

STUDY DESIGN:
Intervention Model Description: Subjects participate in 6 experiments, 3 for each treatment (Elagolix OR Estradiol and placebo). The order of treatment is random.
Who Masked: Participant, Investigator
Masking Description: Double (participant, investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Premenopausal estrogen suppression (Experimental): Participants take a cellulose placebo tablet for 4 days prior to baseline testing and continue until experimental visits are complete. Following completion of placebo testing, participants begin taking 400 mg/day Elagolix for 4 days prior to testing and continue until experimental visits are complete.
  Interventions: Drug: Elagolix Oral Tablet; Other: cellulose placebo
- Postmenopausal estrogen supplementation (Experimental): Participants wear a transdermal estradiol patch or placebo patch for 5 days prior to testing and continue until experimental visits are complete. After 48 hr washout, participants then wear the alternative treatment for 5 days prior to testing until experimental visits are complete.
  Interventions: Drug: Estradiol patch; Other: placebo patch

INTERVENTIONS:
Drug: Elagolix Oral Tablet — 2 x 200 mg tablet
  Other Names: Orilissa
  Arms: Premenopausal estrogen suppression
Drug: Estradiol patch — 0.05 mg/day patch
  Arms: Postmenopausal estrogen supplementation
Other: cellulose placebo — placebo tablet
  Arms: Premenopausal estrogen suppression
Other: placebo patch — placebo patch
  Arms: Postmenopausal estrogen supplementation

SUMMARY:
The frequency and severity of heat waves has increased in the last decades. Older adults (over 65 years) have impaired responses to heat stress making them at increased risk for adverse events. Previous heat waves report that women over 65 experience worse health outcomes than any other age group and age matched men.

Aging and reproductive hormones, specifically estrogen, independently alter responses to heat stress. However, the combined effects of low estrogen following menopause and aging on the response to heat stress are unknown. In this study, the investigators will identify the role of estrogen in pre and post menopausal women on thermoregulatory responses to heat stress.

DETAILED DESCRIPTION:
Premenopausal and postmenopausal women will be recruited and different interventions will be given to each group. To mimic a postmenopausal hormone profile, premenopausal women will be given a GnRH antagonist, which acutely reduces estrogen concentrations. This induces a temporary post-menopausal state without compounding aging effects. Postmenopausal women will be given a transdermal estradiol patch to acutely raise estrogen concentrations. Supplementing estrogen in postmenopausal women allows for the effect of menopausal low estrogen concentration to be removed from the physiological effects of aging.

Subjects sign an informed consent form and undergo a medical screening prior to participation. The screening includes a physical exam, anthropometry, chemical and lipid profiles.

Each subject will complete 6 (3 for each treatment) experimental trials. For each intervention, participants will complete one passive heating experiment first, followed by two active heating experiments.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 42-64

Exclusion Criteria:

* Chron's disease, diverticulitis, or similar gastrointestinal disease
* Abnormal resting exercise electrocardiogram (ECG)
* Tobacco use
* High-risk determined by the Atherosclerotic Cardiovascular Disease (CVD) Risk Factor
* Assessment
* Using hormone therapy
* Using hormonal contraceptives

Ages: 42 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Skin Blood Flow | Monitored continuously during both 3 hour passive heating experiments (Visit 1 and Visit 3 approx 3 weeks)
  Skin blood flow response to whole body heating is continuously monitored
Local Sweat Rate | Monitored continuously during both 3 hour passive heating experiments (Visit 1 and Visit 3 approx 3 weeks)
  A small sweat capsule is placed on the forearm for the duration of whole body heating.
Core Temperature | Monitored continuously during all 3 hour experimental visits (6 total average of 3 weeks)
  Changes in body temperature are measured through a telemetry pill swallowed before each experiment.

SECONDARY OUTCOMES:
Body Mass | Baseline and following 3 hr experimental visit (6 total visits for study completion, an average of 3 weeks)
  Body mass is measured on a scale.
Skin Temperature | Calculated continuously for the duration of each 3 hr experimental visit (6 total visits for study completion, an average of 3 weeks)
  Mean skin temperature is calculated from a weighted average of skin temperature from 4 different sites.

CONTACTS AND LOCATIONS:
Overall Officials: W. Larry Kenney, Ph.D., Principal Investigator — The Pennsylvania State University
Locations (1):
- Noll Laboratory, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No